CLINICAL TRIAL: NCT02410967
Title: Attention Bias Modification Training in Youth With Subthreshold Impairing Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UH2MH101470 (NIH)
Record Dates: First submitted 2015-03-17; First posted 2015-04-08 (Estimated); Results first posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-05

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Attention Bias Modification (Experimental): Attention Bias Modification is a computer-based attention training program.
  Interventions: Behavioral: Attention Bias Modification
- Placebo Attention Task (Placebo Comparator): The Placebo Attention Task uses the same computer-based format and stimuli as the Attention Bias Modification Task, but does not train attention toward or away from stimuli.
  Interventions: Behavioral: Placebo Attention Task

INTERVENTIONS:
Behavioral: Attention Bias Modification — At each of eight sessions, participants complete 160 computer administered trials wherein a pair of threatening stimuli and neutral stimuli is presented simultaneously and then followed immediately by a probe. The probe always replaces the neutral stimulus and never replaces the threatening stimulus. The intervention is based on the idea that attention can be shaped via repetitive computer based training methods, and training attention toward neutral stimuli will lead to a reduction in anxiety and its disorders.
  Arms: Attention Bias Modification
Behavioral: Placebo Attention Task — At each of eight sessions, participants complete 160 computer administered trials wherein a pair of threatening stimuli and neutral stimuli is presented simultaneously and then followed immediately by a probe. The probe replaces the neutral stimulus and the threatening stimulus with equal probability.
  Arms: Placebo Attention Task

SUMMARY:
This study is a pilot test of Attention Bias Modification Training (ABMT) among clinic referred children and adolescents with subthreshold impairing anxiety (i.e., anxiety and related impairment that fails to meet criteria for an anxiety disorder diagnosis). Half of participants will receive 8 sessions of computer administered ABMT and the other half of participants will receive a 8 sessions of a computer administered control task.

DETAILED DESCRIPTION:
This study will collect preliminary data on Attention Bias Modification Training (ABMT) among clinic referred children and adolescents who display subthreshold impairing anxiety (SubImpAnx; anxiety & related impairment that fails to meet diagnostic criteria for an anxiety disorder). Traditional approaches to mental health service delivery cannot meet current demand. The inadequacies of traditional service delivery are magnified when viewed through the lens of impaired but undiagnosed youth. It is an unaddressed empirical question whether a least restrictive treatment can effectively reduce SubImpAnx in youth. Empirical efforts to address this issue are important because youths with SubImpAnx experience substantial impairment, are at high risk of escalation to full syndrome anxiety disorder, and pose a burden on the health care system.

This study will enroll 66 clinic referred children and adolescents (ages 8-16 years) who meet criteria for SubImpAnx. Participants will be randomly assigned to complete 8 sessions of either ABMT or a placebo control (PC) task over 4 weeks. Clinician ratings on youth anxiety severity and impairment will be evaluated as the primary outcome. Youth self ratings and parent ratings on youth anxiety symptoms and impairment will be evaluated as secondary outcomes. All measures will be collected before condition assignment (pretreatment), at immediate posttreatment, and at an 8 week follow up. In addition, initial data will be collected to shed light on whether it would be useful to pursue (a) attention bias to threat as a mediator of ABMT's anxiety reduction effects and (b) dose-response issues related to ABMT's anxiety reduction effects in a subsequent, larger study.

The specific aims are: Collect pilot data on the effects of ABMT and a PC task on levels of anxiety and impairment at a post evaluation (Aim 1) and at a follow up (FU) evaluation 8 weeks after the post evaluation (Aim 2); Preliminarily examine whether ABMT leads to lower levels of attention bias toward threatening stimuli as compared to a PC Task at post and 8 week FU (Aim 3); Describe the course of anxiety symptoms and impairment during treatment among youth in the ABMT condition (Aim 4).

This project will provide critically needed pilot data on ABMT for youth with SubImpAnx. With these data in hand, the field will be in a better position to determine whether ABMT may be used as a least restrictive intervention among anxious youth who are 'impaired but undiagnosed.'

ELIGIBILITY:
Inclusion Criteria:

* 8-16 years old
* meet criteria for subthreshold impairing anxiety

Exclusion Criteria:

* meet diagnostic criteria for Anxiety Disorder, Organic Mental Disorders, Psychotic Disorders, Pervasive Developmental Disorders, or Mental Retardation
* a high likelihood of harming self or others
* not been living with a primary caregiver for at least 6 months who is legally able to give consent for the child's participation
* previously undisclosed abuse requiring investigation or ongoing supervision by the Department of Social Services;
* involved currently in another psychosocial/behavioral treatment
* a serious vision problem that is not corrected with prescription lenses
* a physical disability that interferes with the ability to click a mouse button rapidly and repeatedly

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2014-07; Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Pettit, PhD, Principal Investigator — Florida International University
Locations (1):
- Florida International University Center for Children and Families, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Trial Period: Treatment Phase (4 Weeks) Total Started: 53 [Protocol Enrollment: 53]
  Trial Period:Follow-up Phase (8 Weeks) Total Started: 48
Period: Treatment Phase (4 Weeks)
Arm/Group | Attention Bias Modification | Placebo Attention Task
Started | 27 | 26
Completed | 26 | 22
Not Completed | 1 | 4
Period: Follow-up Phase (8 Weeks)
Arm/Group | Attention Bias Modification | Placebo Attention Task
Started | 26 | 22
Completed | 22 | 16
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Attention Bias Modification | Placebo Attention Task | Total
Number analyzed (Participants) | 27 | 26 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 27 | 26 | 53
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.67 (2.68) | 8.85 (2.53) | 9.27 (2.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 17 | 12 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 16 | 35
  Not Hispanic or Latino | 6 | 10 | 16
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 26 | 21 | 47
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27 | 26 | 53

OUTCOME MEASURES:

1. Primary Outcome: Pediatric Anxiety Rating Scale at Posttreatment
Description: posttreatment clinician rating of youth anxiety symptom severity over the past 7 days. The name of the measure is the Pediatric Anxiety Rating Scale (PARS). The PARS is a clinician rated measure of the severity of youths' anxiety symptoms. Total scores on the PARS range from 0 to 35, with higher scores representing more severe anxiety.
Time Frame: 7 days
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Attention Bias Modification | Placebo Attention Task
Number analyzed (Participants) | 27 | 26
units on a scale | 7.21 (5.66) | 7.73 (4.81)

2. Primary Outcome: Pediatric Anxiety Rating Scale at Follow-up
Description: follow-up clinician rating of youth anxiety symptom severity over the past 7 days. The name of the measure is the Pediatric Anxiety Rating Scale (PARS). The PARS is a clinician rated measure of the severity of youths' anxiety symptoms. Total scores on the PARS range from 0 to 35, with higher scores representing more severe anxiety.
Time Frame: 7 days
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Attention Bias Modification | Placebo Attention Task
Number analyzed (Participants) | 27 | 26
units on a scale | 8.42 (6.21) | 5.69 (4.42)

3. Secondary Outcome: Screen for Child Anxiety Related Emotional Disorders - Parent Version at Posttreatment
Description: posttreatment parent rating of youth anxiety symptom severity over the past 14 days. The name of the measure is the Screen for Child Anxiety Related Emotional Disorders - Parent Version (SCARED-P). The SCARED-P is a parent rated measure of the severity of youths' anxiety symptoms. Total scores on the SCARED-P range from 0 to 82, with higher scores representing more severe anxiety.
Time Frame: 14 days
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Attention Bias Modification | Placebo Attention Task
Number analyzed (Participants) | 27 | 26
units on a scale | 19.82 (14.54) | 20.16 (11.75)

4. Secondary Outcome: Screen for Child Anxiety Related Emotional Disorders - Parent Version at Follow-up
Description: follow-up parent rating of youth anxiety symptom severity over the past 14 days. The name of the measure is the Screen for Child Anxiety Related Emotional Disorders - Parent Version (SCARED-P). The SCARED-P is a parent rated measure of the severity of youths' anxiety symptoms. Total scores on the SCARED-P range from 0 to 82, with higher scores representing more severe anxiety.
Time Frame: 14 days
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Attention Bias Modification | Placebo Attention Task
Number analyzed (Participants) | 27 | 26
units on a scale | 21.96 (16.82) | 17.13 (10.86)

5. Secondary Outcome: Screen for Child Anxiety Related Emotional Disorders - Child Version at Posttreatment
Description: posttreatment youth self-rating of youth anxiety symptom severity over the past 14 days. The name of the measure is the Screen for Child Anxiety Related Emotional Disorders - Child Version (SCARED-C). The SCARED-C is a child self-rated measure of the severity of youths' anxiety symptoms. Total scores on the SCARED-C range from 0 to 82, with higher scores representing more severe anxiety.
Time Frame: 14 days
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Attention Bias Modification | Placebo Attention Task
Number analyzed (Participants) | 27 | 26
units on a scale | 17.88 (13.76) | 14.72 (10.61)

6. Secondary Outcome: Screen for Child Anxiety Related Emotional Disorders - Child Version at Follow-up
Description: follow-up youth self-rating of youth anxiety symptom severity over the past 14 days. The name of the measure is the Screen for Child Anxiety Related Emotional Disorders - Child Version (SCARED-C). The SCARED-C is a child self-rated measure of the severity of youths' anxiety symptoms. Total scores on the SCARED-C range from 0 to 82, with higher scores representing more severe anxiety.
Time Frame: 14 days
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Attention Bias Modification | Placebo Attention Task
Number analyzed (Participants) | 27 | 26
units on a scale | 20.41 (15.66) | 11.88 (10.88)

ADVERSE EVENTS:
Time Frame: 3-month time period from pre-treatment evaluation to 2-month follow-up evaluation
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign, symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Attention Bias Modification | Placebo Attention Task
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/26
Other Adverse Events (participants affected / at risk) | 0/27 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/67/NCT02410967/Prot_SAP_000.pdf